CLINICAL TRIAL: NCT01006473
Title: A Randomized Trial of the Effects of Exercise Training in Chagas Cardiomyopathy
Brief Title: Exercise Training in Chagas Cardiomyopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Antonio Luiz Pinho Ribeiro, Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNPq402024/2005-2
Record Dates: First submitted 2009-11-01; First posted 2009-11-02 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Chagas Disease; Cardiomyopathy; Exercise Training
Keywords: Chagas Disease; Chagas Cardiomyopathy; Exercise Movement Techniques
MeSH Terms: conditions — Chagas Disease; Cardiomyopathies; Chagas Cardiomyopathy | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise training group (Experimental): Exercise training is performed in subgroups of 6 patients supervised by two physiotherapists. Exercise prescription consisted of a 15-min warm-up, walking up to 30 min, followed by a 15-min cooling-down. The exercise intensity during the first 2 weeks corresponds to 55% at 65% of the HR peak reached at the baseline exercise test. In posterior sessions, individual adjustments are performed with gradual increases in order to reach the adequate target HR training intensity, as determined by the Karvonen formula {(maximal HR - HR at rest) x 50 to 70% + HR at rest}. Exercise training is performed in the morning, three times a week (on alternate days) for a total of 12 weeks (36 sessions).
  Interventions: Other: Exercise training
- Inactive control group (No Intervention): No intervention

INTERVENTIONS:
Other: Exercise training
  Arms: Exercise training group

SUMMARY:
The benefits of exercise training in heart failure are well established. Its effects, however, have not been evaluated in Chagas cardiomyopathy (ChC). The investigators hypothesis is that the exercise training may improve functional capacity, quality of life (QoL), and reduce brain natriuretic peptide (BNP) levels in patients with ChC.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Chagas dilated cardiomyopathy, defined by the echocardiography finding of a dilated left ventricle with moderate or severe impaired left ventricular systolic function (left ventricular ejection fraction ≤ 45%).
* To be clinically stable for at least 3 months
* To have sinus rhythm
* To be under standard medical therapy use at the time.

Exclusion Criteria:

* Inability to attend regular exercise training
* The presence of a pacemaker, associated cardiac or systemic diseases
* Practitioners of regular physical activity

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Functional capacity | 12 weeks
Functional class | 12 weeks
Health related quality of life | 12 weeks
BNP levels | 12 weeks

SECONDARY OUTCOMES:
Complications related to the exercise training | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antonio L Ribeiro, MD, PhD, Study Chair — Federal University of Minas Gerais; Manoel Otávio C Rocha, MD, PhD, Principal Investigator — Federal University if Minas Gerais; Maria do Carmo P Nunes, MD, PhD, Study Director — Federal University of Minas Gerais
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Result] Lima MM, Rocha MO, Nunes MC, Sousa L, Costa HS, Alencar MC, Britto RR, Ribeiro AL. A randomized trial of the effects of exercise training in Chagas cardiomyopathy. Eur J Heart Fail. 2010 Aug;12(8):866-73. doi: 10.1093/eurjhf/hfq123. PMID 20675669
- [Result] Lima MM, Nunes MC, Nascimento B, Costa HS, Sousa LA, Teixeira AL, Rocha MO, Ribeiro AL. Improvement of the functional capacity is associated with BDNF and autonomic modulation in Chagas disease. Int J Cardiol. 2013 Sep 1;167(5):2363-6. doi: 10.1016/j.ijcard.2012.11.055. Epub 2012 Dec 8. No abstract available. PMID 23232458
- [Result] Lima MM, Nunes MC, Rocha MO, Beloti FR, Alencar MC, Ribeiro AL. Left ventricular diastolic function and exercise capacity in patients with Chagas cardiomyopathy. Echocardiography. 2010 May;27(5):519-24. doi: 10.1111/j.1540-8175.2009.01081.x. Epub 2010 Apr 16. PMID 20412275
- [Result] Nascimento BR, Lima MM, Nunes Mdo C, Alencar MC, Costa HS, Pinto Filho MM, Cota VE, Rocha MO, Ribeiro AL. Effects of exercise training on heart rate variability in Chagas heart disease. Arq Bras Cardiol. 2014 Sep;103(3):201-8. doi: 10.5935/abc.20140108. Epub 2014 Aug 1. PMID 25098373